CLINICAL TRIAL: NCT03184324
Title: A Multi-Center, Randomized, Double-Blind, Active-controlled, Phase 2, Therapeutic Exploratory Study to Evaluate the Efficacy and Safety of DWP14012 in Patients With Erosive Gastroesophageal Reflux Disease.
Brief Title: Study to Evaluate the Efficacy and Safety of DWP14012 in Patients With Erosive Gastroesophageal Reflux Disease (Phase 2, Therapeutic Exploratory Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP14012002
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2018-06

CONDITIONS: Erosive Gastroesophageal Reflux Disease
MeSH Terms: interventions — fexuprazan; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DWP14012 20mg (Experimental): DWP14012 20mg, tablet, orally, once daily
  Interventions: Drug: DWP14012; Drug: DWP14012 placebo; Drug: Esomeprazole placebo
- DWP14012 40mg (Experimental): DWP14012 40mg, tablet, orally, once daily
  Interventions: Drug: DWP14012; Drug: DWP14012 placebo; Drug: Esomeprazole placebo
- DWP14012 80mg (Experimental): DWP14012 40mg*2, tablet, orally, once daily
  Interventions: Drug: DWP14012; Drug: DWP14012 placebo; Drug: Esomeprazole placebo
- Esomerpazole 40mg (Active Comparator): Esomerpazole 40mg, tablet, orally, once daily
  Interventions: Drug: Esomeprazole; Drug: DWP14012 placebo

INTERVENTIONS:
Drug: DWP14012 — tablet
  Arms: DWP14012 20mg; DWP14012 40mg; DWP14012 80mg
Drug: Esomeprazole — tablet
  Other Names: Nexium
  Arms: Esomerpazole 40mg
Drug: DWP14012 placebo — tablet
Drug: Esomeprazole placebo — tablet
  Arms: DWP14012 20mg; DWP14012 40mg; DWP14012 80mg

SUMMARY:
The purpose of this study is to determine the efficacy and safety of DWP14012 compared to esomeprazole in the treatment of erosive gastroesophageal reflux disease classified as Los Angeles(LA) classification grades A to D.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 20 and 75 years old based on the date of written agreement
* Those who have been diagnosed with erosive gastroesophageal reflux disease(EGRD) of LA Grade A-D on the upper gastrointestinal endoscopy
* Those who experienced symptoms of heartburn or acid reflux within the last 7 days

Exclusion Criteria:

* Those who have undergone gastric acid suppression or gastric, esophageal surgery
* Those who with clinically significant liver, kidney, nervous system, respiratory, endocrine, hematologic, cardiovascular, urinary system disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Ratio of subjects who were completely cured of mucosal defects by 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Ratio of subjects who were completely cured of mucosal defects by 4 weeks | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Medical Center, Sungdong-gu, Seoul, South Korea